CLINICAL TRIAL: NCT04106466
Title: Deep Brain Stimulation (DBS) for Treatment Resistant Depression: Exploration of Local Field Potentials (LFPs) With the Medtronic Summit RC+S "Brain Radio" System
Brief Title: DBS for TRD With the Medtronic Summit RC+S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Mayberg, MD (Other)
Collaborators: Emory University (Other); Georgia Institute of Technology (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Helen Mayberg, MD, Professor, Departments of Neurology, Neurosurgery, Neuroscience, Psychiatry, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 17-2763; 5UH3NS103550 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Deep Brain Stimulation; Major Depressive Disorder; Treatment resistant depression; subcallosal cingulate white matter; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Intervention Model Description: All participants will be implanted with the study device and receive open label, active DBS stimulation
Masking Description: N/A. This is open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Deep Brain Stimulation (DBS) (Experimental): Open label active Deep Brain Stimulation (DBS)
  Interventions: Device: Medtronic Summit RC+S DBS system

INTERVENTIONS:
Device: Medtronic Summit RC+S DBS system — Open label active Deep Brain Stimulation (DBS)

SUMMARY:
Of the estimated 30 million Americans who suffer from Major Depressive Disorder, approximately 10% are considered treatment resistant. Deep brain stimulation (DBS) to a region of the brain called the subcallosal cingulate (SCC) is an emerging strategy for treatment resistant depression (TRD), which involves placement of electrodes in a specific region of the brain and stimulating that area with electricity. This is believed to reset the brain network responsible for symptoms and results in a significant antidepressant response. A series of open-label studies have demonstrated sustained, long-term antidepressant effects in 40-60% of patients who received this treatment. A challenge to the effective dissemination of this fledgling treatment is the absence of biomarkers (objective, measureable indications of the state of the body and brain) to guide device placement and select stimulation parameters during follow-up care.

By using an experimental prototype DBS device called the Summit RC+S (Medtronic, Inc) which has the ability to both deliver stimulation to and record electrical signals directly from the brain, this study aims to identify changes in local field potentials (LFPs), specific electrical signals that are thought to represent how the brain communicates information from one region to another, to see how this relates to DBS parameter settings and patient depressive symptomatology. The goal of this study is to study LFPs before and during active DBS stimulation to identify changes that correlate with the antidepressant effects of SCC DBS.

The study team will recruit 10 patients with TRD and implant them with the Summit RC+S system. Participants will be asked to complete short questionnaires and collect LFP data twice daily for the first year of the study, as well as have weekly in person research procedures and assessments with the study team for up to one year. These include meetings with the study psychiatrist, psychologist, symptom ratings, and periodic EEGs (scalp brainwave recordings). A brief discontinuation experiment will be conducted after 6 months of stimulation, in which the device will be turned off and patterns of LFP changes will be recorded. The entire study is expected to last about 10 years, which is the expected life of the battery that powers the device. All participants are required to live in the New York metropolitan area for the first two years of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70 years old.
* Ability to provide written informed consent.
* Lives within commuting distance to New York City and study location (Mount Sinai West Hospital)
* Primary psychiatric diagnosis of Major Depressive Disorder (MDD), either single episode or recurrent type, without psychotic features, currently experiencing a Major Depressive Episode (MDE), as diagnosed by Structured Clinical Interview for DSM IV-TR (SCID). Two independent psychiatrists will confirm the diagnosis.
* Current depressive episode of at least two years duration OR a history of more than 3 lifetime depressive episodes.
* Minimum score at study entry of 20 on the 17-item Hamilton Depression Rating Scale (HDRS-17)
* Average pre-operative HDRS-17 score of 20 or greater (averaged over four weekly pre-surgical evaluations during the four weeks prior to surgery) and an average pre-operative HDRS-17 score no more than 30% lower than the baseline screening HDRS-17 score.
* A maximum Global Assessment of Functioning of 50 or less.
* Confirmed to have treatment-resistant depression (TRD). Treatment-resistance will be defined as:

  1. Failure to respond to a minimum of four different antidepressant treatments (including at least three medications from at least three different drug classes), evidence-based psychotherapy, or electroconvulsive therapy (ECT) administered at adequate doses and duration during the current episode. We will require documentation (i.e., statement from the treating psychiatrist) that a treatment trial has failed (either no response to maximum tolerable doses for a minimum of 4 weeks, or side effects at sub-maximal doses) as coded by a revised Antidepressant Treatment History Form (ATHF). The study investigators will confirm each treatment via review of records from referring psychiatrists and/or pharmacy records.
  2. Failure or intolerance of an adequate course of electroconvulsive therapy (ECT) during any episode (confirmed by medical records) or not receiving ECT due to a reason considered valid by the study psychiatrist. Such reasons might include lack of availability of ECT providers in the patient's location, concern regarding the impact of cognitive side effects of ECT on current ability to work or function, or inability to obtain third-party payment for ECT. Additionally, it is recognized that the probability that a patient who has failed four medications in the current episode will achieve a lasting response with ECT is about 18% (60% probability of an acute response and 30% of maintaining response for at least 24 weeks); patients who have refused ECT because they feel the chance of benefit does not outweigh the risks associated with ECT will be considered eligible.
* Able to undergo preoperative MRI
* Have a designated caregiver available to assist in compliance with study procedures
* Willing and able to comply with all study-related appointments and procedures

Exclusion criteria:

* Other Axis I comorbid conditions
* Active suicidal ideation with intent, suicide attempt within the last six months, more than three suicide attempts within the last two years, or serious suicide risk as determined by the study psychiatrists
* Other primary neurological disorders or unstable medical illness
* Conditions requiring anticoagulant therapy which cannot be discontinued for the perioperative period, as required
* Conditions requiring MRI scans or diathermy
* Pregnancy or plan to come pregnant during the study
* Contraindications for general anesthesia, neurosurgery, or an MRI scan
* Currently implanted with a cardiac pacemaker / defibrillator or other implanted electrical device which may interfere with DBS stimulator or the function of which may be impacted by its implantation.
* Patients who lack the capacity for proper device usage and maintenance, in the opinion of the research team

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS) score | Baseline; after 6 months of continuous active stimulation; after 1 year of continuous active stimulation
  Change in Hamilton Depression Rating Scale (HDRS) score at 6 months and 1 year of continuous active stimulation as compared to preoperative baseline. The score for Hamilton Depression Rating Scale, 17 item version, full range from 0-50, with a higher score indicating more severe depression.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline; after 6 months of continuous active stimulation; after 1 year of continuous active stimulation
  Change in Montgomery-Asberg Depression Rating Scale (MADRS) after 6 months and 1 year of continuous active stimulation compared to baseline. MADRS items are rated on a 0 to 6 continuum (0 = no abnormality, 6 = severe). Total score range from 0 to 60, with higher total scores indicating increased severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mayberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (learned intermediary) identified for this purpose may request access to individual participant data meta-analysis. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (https://dabi.loni.usc.edu).
URL: https://dabi.loni.usc.edu

REFERENCES:
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, Crowell AL, Garlow SJ, Rajendra JK, McIntyre CC, Gross RE, Mayberg HS. A connectomic approach for subcallosal cingulate deep brain stimulation surgery: prospective targeting in treatment-resistant depression. Mol Psychiatry. 2018 Apr;23(4):843-849. doi: 10.1038/mp.2017.59. Epub 2017 Apr 11. PMID 28397839
- [Background] Waters AC, Veerakumar A, Choi KS, Howell B, Tiruvadi V, Bijanki KR, Crowell A, Riva-Posse P, Mayberg HS. Test-retest reliability of a stimulation-locked evoked response to deep brain stimulation in subcallosal cingulate for treatment resistant depression. Hum Brain Mapp. 2018 Dec;39(12):4844-4856. doi: 10.1002/hbm.24327. Epub 2018 Aug 18. PMID 30120851
- [Background] Riva-Posse P, Holtzheimer PE, Garlow SJ, Mayberg HS. Practical considerations in the development and refinement of subcallosal cingulate white matter deep brain stimulation for treatment-resistant depression. World Neurosurg. 2013 Sep-Oct;80(3-4):S27.e25-34. doi: 10.1016/j.wneu.2012.11.074. Epub 2012 Dec 13. PMID 23246630
- [Background] Crowell AL, Garlow SJ, Riva-Posse P, Mayberg HS. Characterizing the therapeutic response to deep brain stimulation for treatment-resistant depression: a single center long-term perspective. Front Integr Neurosci. 2015 Jun 15;9:41. doi: 10.3389/fnint.2015.00041. eCollection 2015. PMID 26124710
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, McIntyre CC, Gross RE, Chaturvedi A, Crowell AL, Garlow SJ, Rajendra JK, Mayberg HS. Defining critical white matter pathways mediating successful subcallosal cingulate deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2014 Dec 15;76(12):963-9. doi: 10.1016/j.biopsych.2014.03.029. Epub 2014 Apr 13. PMID 24832866

DOCUMENTS (1):
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT04106466/ICF_000.pdf